CLINICAL TRIAL: NCT00017342
Title: Phase II Study Of Bryostatin 1 (NSC 339555) And High-Dose 1-B-D-Arabinofuranosylcytosine (HiDAC) In Patients With Refractory Leukemia
Brief Title: Bryostatin 1 and Cytarabine in Treating Patients With Relapsed Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven Grant, MD, Virginia Commonwealth University
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068679; P30CA016059 (NIH); MCV-MCC-4710; NCI-4710
Record Dates: First submitted 2001-06-06; First posted 2003-02-06 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — bryostatin 1; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1
Drug: cytarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining bryostatin 1 with cytarabine in treating patients who have relapsed primary acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with primary acute myelogenous leukemia in first relapse treated with bryostatin 1 and high-dose cytarabine.
* Determine the toxic effects of this regimen in these patients.
* Determine the relapse-free survival and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction: Patients receive bryostatin 1 IV over 24 hours on days 1 and 11. Patients also receive high-dose cytarabine IV over 3 hours every 12 hours for 4 infusions on days 2-3 and days 9-10.

Patients who achieve a major response receive a second course of induction therapy.

* Consolidation: Patients who achieve complete remission receive bryostatin 1 IV over 24 hours on days 1 and 10 and high-dose cytarabine IV over 3 hours every 12 hours for 2 infusions on days 2 and 9. Treatment continues for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients who achieve a response and subsequently relapse may receive additional induction and consolidation therapy at the discretion of the investigator.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 15-46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary acute myelogenous leukemia (AML) in first relapse after a remission of at least 3 months duration
* No secondary AML, including the following:

  * Therapy-related AML
  * AML arising from myelodysplastic syndromes or similar hematological conditions
* No Philadelphia chromosome or other evidence of a (9;21) translocation
* Ineligible for potentially curative allogeneic stem cell transplantation

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (patients with Gilbert's disease or unconjugated hyperbilirubinemia may have bilirubin no greater than 3.0 mg/dL with conjugated bilirubin no greater than 0.5 mg/dL)
* AST/ALT no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Pulmonary:

* No clinically significant pulmonary disease

Other:

* No clinically significant cytarabine-related cerebellar toxicity
* No nonmalignant systemic disease that causes poor medical risk
* No active, uncontrolled, serious infection
* No medical condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior allogeneic stem cell transplantation

Chemotherapy:

* At least 2 weeks since prior systemic chemotherapy (24 hours for hydroxyurea) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Recovered from all prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2004-09 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, MD, Study Chair — Massey Cancer Center
Locations (4):
- United States (4):
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia